CLINICAL TRIAL: NCT05477238
Title: Oxygen Consumption in Post-stroke Patients During Various Walking Activities Compared to Healthy Controls
Acronym: STROXCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 87RI22_0005 (STROXCO)
Record Dates: First submitted 2022-06-23; First posted 2022-07-28 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Cerebrovascular Accident
Keywords: Stroke; Oxygen consumption; physical activity
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Intervention Model Description: Monocentric, cross-sectional and comparative study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cerebrovascular Accident (Experimental): Stroke patients will perform 2 walking tests indoors and outdoors wearing a gas exchange analyzer, an accelerometer and a heart rate monitor meter
  Interventions: Procedure: walking tasks
- healthy volunteer (Other): Healthy volunteers patients will perform 2 walking tests indoors and outdoors wearing a gas exchange analyzer, an accelerometer and a heart rate monitor meter
  Interventions: Procedure: walking tasks

INTERVENTIONS:
Procedure: walking tasks — The experiment will be divided in two sessions. In the first session, the participant/healthy volunteers will do 3 walking tasks (over ground walking/ climbing up, down stairs). In the second session, the participant will walk outside in front of the hospital (walking on a slope, walking down, walking on uneven ground). All those tasks will be done while wearing a gas exchange analyzer, accelerometer and a heart rate meter.

SUMMARY:
Stroke is major public health issue. The investigators recommend post-stroke patients to practice physical activity. Nevertheless, the recommendations are not widely respected due to the intensity of exercises. Oxygen consumption is a parameter to assess the intensity of physical activity. in this sense, we want to measure the oxygen consumption during various walking tasks compared to healthy controls.

DETAILED DESCRIPTION:
Stroke is defined as an interruption of blood circulation in the brain. The treatments are in first time medical in emergency. Then, the patient will start his rehabilitation with several contributors. At this time, it will recommend physical activity to patients. Regardless of the all benefits of physical activity, it will help patient to avoid a second stroke. The investigators have the recommendations of the high authority of health in physical activity for stroke population. It recommends to practice around 20 to 60 minutes daily of physical activity with moderate effort intensity. Oxygen consumption is a parameter of effort intensity of physical activity measured in ml O2/kg/min. Currently, the investigators have the compendium of physical activity (PA). it allows us to classify PA according to effort intensity. And so, an activity with a moderate effort intensity is an activity between 3 and 5.9 metabolic equivalent task (MET). Note that 1 MET is 3.5 ml/O2/Kg. Nevertheless, this compendium does not correspond to post-stroke individuals. As consequences, Low intensity exercise as described in guidelines might be at a moderate intensity level for stroke survivors. Hence, the investigators want to assess the oxygen consumption of post-stroke individuals during various walking tasks and compare it to healthy controls.

ELIGIBILITY:
Inclusion Criteria:

Common to both groups:

* Age >=18 years
* Able to give consent
* Not under guardianship or curatorship
* Enrolled in the French social security system

Specific to the cerebrovascular accident Group:

* Stroke confirmed by brain imaging
* Able to walk stairs without human assistance (modified Functional Ambulation Classification >= 6)

Healthy Group Specific:

- Individuals matched to stroke individuals on age sex and BMI.

Exclusion Criteria:

Cerebrovascular accident group - Severe cognitive impairment (MoCA < 18)

Common to both groups:

- Presence of contraindication to physical activity: unstable diabetes, unstable hypertension, unstable angina, intra-cardiac thrombus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Oxygen consumption measurement | Day 1
  Oxygen consumption by indirect calorimetry (respiratory gas exchange analyzer: Metamax) expressed in mL.min-1.kg-1
Oxygen consumption measurement | Day 7
  Oxygen consumption by indirect calorimetry (respiratory gas exchange analyzer: Metamax) expressed in mL.min-1.kg-1

SECONDARY OUTCOMES:
Walking speed measurement | Day 1
  Average walking speed measured (distance walked/total time) during different travel activities
Walking speed measurement | Day 7
  Average walking speed measured (distance walked/total time) during different travel activities
Cardiac frequency measurement | Day 1
  Average heart rate during activity measured by heart rate meter in bpm
Cardiac frequency measurement | Day 7
  Average heart rate during activity measured by heart rate meter in bpm
Perception of effort | Day 1
  Perception of effort by the Borg scale during the last minute of the movement activity
Perception of effort | Day 7
  Perception of effort by the Borg scale during the last minute of the movement activity
Total energy expenditure | Day 1
  Total energy expenditure during each movement activity estimated by an Actigraph GT3X placed at the healthy ankle
Total energy expenditure | Day 7
  Total energy expenditure during each movement activity estimated by an Actigraph GT3X placed at the healthy ankle

CONTACTS AND LOCATIONS:
Locations (1):
- Limoges university hospital, Limoges, France